CLINICAL TRIAL: NCT03278353
Title: The Mediating Effect of Baseline Expectations of Conservative Care and Surgery Outcomes on Fulfillment of Expectations for Patients With Femoroacetabular Impingement Syndrome
Brief Title: Fulfillment of Expectations for Patients With FAI Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00084795
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Femoroacetabular Impingement
Keywords: Expectation; Conservative Intervention
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Prospective cases series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conservative care (Experimental): Exercise and manual therapy
  Interventions: Other: Exercise; Other: Manual Therapy

INTERVENTIONS:
Other: Exercise — A prescription of progressive rehabilitation exercises designed to strengthen weakened muscle groups and stretch joint movements that demonstrate range of motion limitations will be provided as a home program. Treatment is based on clinical presentation and identification of impairments by the treating clinician. Participants will be seen for 3 visits over 6 weeks and a final visit 1 year post-surgery for those electing to undergo surgery.
  The interventions will consist of progressive exercise (PE) in two phases with general instruction guidelines. The assigned program will be tailored per each participant's clinical presentation and progressed based on response to exercise load. The researcher will instruct, review and supervise each program initially and, at follow-up visits; as well as monitor progress, re-enforce treatment strategies and modify the respective program accordingly. Each participant will receive a home program manual as well as a program log.
Other: Manual Therapy — Hip joint and spine manual therapy techniques applied toward the impairments of the subject.

SUMMARY:
A total of 63 participants will be recruited through 3 local surgeons in Durham, North Carolina after distinctive differential diagnostic methods, all with extensive expertise in intra-articular hip pathology and arthroscopy. The surgeons will offer the opportunity to participate in the trial by providing information to the recipient. Potential participants that do not contact project team members will be contacted by phone if they do not respond to the initial invitation. Potential participants will be initially screened by telephone interview, followed by a clinical examination to confirm study eligibility. The blinded researchers will obtain informed consent and will perform outcome assessments

Purpose of the Study: 1) measure the mediating effect of baseline patient expectations on fulfillment of expectations (for both conservative care and surgery, measured at 6 weeks and at 1 year respectively) in a cohort of patients with a diagnosis of FAI Syndrome who receive six weeks of conservative physical therapy intervention and 2) measure the effect of baseline expectations on patient reported outcomes (e.g., HAGOS, pain, global rating of change) at six weeks.

DETAILED DESCRIPTION:
FAI Syndrome is a morphological hip condition that can cause hip/groin pain and impaired performance.1 FAI Syndrome is caused by abnormal morphology of the femoral head (referred to as cam FAI Syndrome), excessive acetabular coverage of the femoral head (referred to as pincer FAI Syndrome) or a combination of the two (mixed FAI Syndrome).2 Not only can FAI Syndrome give rise to symptoms and impair function, the repetitive bony contact can also lead to a cascade of structural damage including tearing at the chondrolabral junction, full thickness cartilage delamination, and potentially hip osteoarthritis.

Presently, there is uncertainty involving the best treatment approach for symptomatic FAI Syndrome.2 The principal two management options are 1) physical therapy management of impairments and function and/or 2) surgery. Although presently, both modalities have been shown to improve symptoms in the short term,2 surgery is by far the most commonly incorporated approach.1, The incidence of the surgery has notably increased in recent years. There has been an 18-fold increase in surgical procedures for FAI Syndrome between 1999 and 2009, varying by geographic region in the USA.3

As an elective procedure, surgery for correction of FAI Syndrome is likely influenced by patients' perspectives and expectations of outcome.4 The extent to which these expectations influence specific treatment choices, as well as subsequent outcomes is currently unclear, although recent findings suggest that across various pathologies both patients5 and clinicians6 rarely have accurate expectations of treatment benefits or harms.

Non-operative, conservative treatments may have a role in managing FAI Syndrome to alleviate symptoms, potentially resulting in postponement or avoidance of surgery. Bony morphological changes can be present without symptoms, and nearly all participants with symptomatic FAI Syndrome undergo a variable asymptomatic period in the presence of structural FAI Syndrome. Recent studies have been hampered by retrospective and case cohort design, very small sample sizes, short-term follow up, and self-report measures only.4 A recent systematic review stated "although the available literature with experimental data is limited, there is a suggestion that physical therapy and activity modification confer some benefit to patients. Non-operative treatment regimens, particularly physical therapy, need to be evaluated more extensively and rigorously".6 Further, it is well known that patient expectations can mediate outcomes. Those who have high expectations about the potential benefit of the conservative approach are more likely to experience improvements. Conversely, those who have low expectations are more likely to fail to see improvement.

4. Design & Procedures: Reporting of the study will conform to STROBE guidelines for observational studies. The proposed study is a prospective case series:

1) Patients will receive:

1. A prescription of progressive rehabilitation exercises designed to strengthen weakened muscle groups and stretch joint movements that demonstrate range of motion limitations. Treatment is based on clinical presentation and identification of impairments by the treating clinician.
2. Education on progression of exercise based on scientific exercise progression principle. Participants will be seen for 3 visits over 6 weeks (with weekly contact with the patient via email or phone call) and a final visit 1 year post-surgery for those electing to undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 18 to 60 years,
* diagnosed with FAI by an orthopedic surgeon and exhibiting
* hip/groin symptoms for at least 3 months (symptomatic); and
* signs, symptoms and imaging findings conducive to FAI will be recruited from a surgical practice of an orthopedic surgeon in Durham, North Carolina.

Exclusion Criteria:

* subjects that have radiographic evidence of hip osteoarthritis that is more than mild in severity defined as Tonnis >grade 1 or Kellgren-Lawrence >2;
* have other concurrent injury/conditions that will affect their ability to participate in the rehabilitation program and/or assessment procedures;
* exhibit hip dysplasia (center edge angle <20 degrees on AP radiograph
* are unable to attend a study physiotherapist or participate in the rehabilitation program if randomized to the PT group;
* are unable to understand English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Fulfillment of expectations with conservative care | 6 weeks post study initiation
  fulfillment of expectations after conservative care implemented as by outcome questionnaire 'Fulfillment of expectations'
Fulfillment of expectations with surgery | 1 year post-surgery
  fulfillment of expectations after surgical care implemented as measured by 'Fulfillment of expectations' questionnaire

SECONDARY OUTCOMES:
Change in Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS) | baseline, 6 weeks and 1 year post-surgery
  patient expectations of care
Expectations of conservative care | baseline
  Expectations of conservative care as measured by expectation survey
Change in Expectations of surgery as measured by expectation survey | baseline and 6 weeks
Change in Reasons for surgery | baseline and 6 weeks
  patient reasons on why choosing surgery
Change in Patient Acceptable Symptom State (PASS) | 6 weeks and 1 year post-surgery
  PASS
Change in Numeric pain rating scale (NPRS) | baseline, 2 weeks, 6 weeks and 1 year
Change in Global Rating of Change Score (GRoC) | 2 weeks, 6 weeks and 1 year post-surgery
  GRoC
Change in Hip and Groin Outcome Score (HAGOS) | baseline, 6 weeks and 1 year post-surgery
  Patient reported outcome measure relative to hip and groin pain
Change in Single Leg Squat (Maximum ROM until onset of pain) | baseline, 6 weeks and 1 year post-surgery
  single leg squat performance
Change in Bilateral Squat (Maximum ROM until onset of pain) | baseline, 6 weeks and 1 year post-surgery
  bilateral leg squat performance
Change in Tegner Activity Scale | baseline, 6 weeks and 1 year post-surgery
  Tegner Activity Scale
Change in Adverse events | baseline, 2 weeks, 6 weeks and 1 year post-surgery
  any adverse events encountered

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reiman, DPT, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Orthopaedic Clinic Page Road, Durham, North Carolina
  - Duke Sports Science Institute, Durham, North Carolina
  - Duke Orthopaedic Clinic, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ayeni O, Chu R, Hetaimish B, Nur L, Simunovic N, Farrokhyar F, Bedi A, Bhandari M. A painful squat test provides limited diagnostic utility in CAM-type femoroacetabular impingement. Knee Surg Sports Traumatol Arthrosc. 2014 Apr;22(4):806-11. doi: 10.1007/s00167-013-2668-8. Epub 2013 Sep 26. PMID 24067989
- [Background] Beck M, Leunig M, Parvizi J, Boutier V, Wyss D, Ganz R. Anterior femoroacetabular impingement: part II. Midterm results of surgical treatment. Clin Orthop Relat Res. 2004 Jan;(418):67-73. PMID 15043095
- [Background] Briggs KK, Lysholm J, Tegner Y, Rodkey WG, Kocher MS, Steadman JR. The reliability, validity, and responsiveness of the Lysholm score and Tegner activity scale for anterior cruciate ligament injuries of the knee: 25 years later. Am J Sports Med. 2009 May;37(5):890-7. doi: 10.1177/0363546508330143. Epub 2009 Mar 4. PMID 19261899
- [Background] Cormier S, Lavigne GL, Choiniere M, Rainville P. Expectations predict chronic pain treatment outcomes. Pain. 2016 Feb;157(2):329-338. doi: 10.1097/j.pain.0000000000000379. PMID 26447703
- [Background] Diamond LE, Dobson FL, Bennell KL, Wrigley TV, Hodges PW, Hinman RS. Physical impairments and activity limitations in people with femoroacetabular impingement: a systematic review. Br J Sports Med. 2015 Feb;49(4):230-42. doi: 10.1136/bjsports-2013-093340. Epub 2014 Sep 22. PMID 25246442
- [Background] Hoffmann TC, Del Mar C. Patients' expectations of the benefits and harms of treatments, screening, and tests: a systematic review. JAMA Intern Med. 2015 Feb;175(2):274-86. doi: 10.1001/jamainternmed.2014.6016. PMID 25531451
- [Background] Hoffmann TC, Del Mar C. Clinicians' Expectations of the Benefits and Harms of Treatments, Screening, and Tests: A Systematic Review. JAMA Intern Med. 2017 Mar 1;177(3):407-419. doi: 10.1001/jamainternmed.2016.8254. PMID 28097303
- [Background] Kemp JL, Makdissi M, Schache AG, Pritchard MG, Pollard TC, Crossley KM. Hip chondropathy at arthroscopy: prevalence and relationship to labral pathology, femoroacetabular impingement and patient-reported outcomes. Br J Sports Med. 2014 Jul;48(14):1102-7. doi: 10.1136/bjsports-2013-093312. Epub 2014 Mar 21. PMID 24659505
- [Background] Reiman MP, Thorborg K, Holmich P. Femoroacetabular Impingement Surgery Is on the Rise-But What Is the Next Step? J Orthop Sports Phys Ther. 2016 Jun;46(6):406-8. doi: 10.2519/jospt.2016.0605. PMID 27245488
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Wall PD, Fernandez M, Griffin DR, Foster NE. Nonoperative treatment for femoroacetabular impingement: a systematic review of the literature. PM R. 2013 May;5(5):418-26. doi: 10.1016/j.pmrj.2013.02.005. Epub 2013 Feb 16. PMID 23419746